CLINICAL TRIAL: NCT03547895
Title: Real Life Experience in the Management of HCV Related Decompensated Cirrhosis With Direct Antiviral Agents
Brief Title: Management of Decompensated HCV Cirrhotic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Amr Shaaban Hanafy, Assistant professor, Zagazig University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3778
Record Dates: First submitted 2017-05-27; First posted 2018-06-06 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Decompensated Cirrhosis
MeSH Terms: interventions — Sofosbuvir; daclatasvir; Ribavirin; Vitamin K; Vitamin K 1; Furosemide; Spironolactone; milk-thistle extract; Silymarin

STUDY DESIGN:
Intervention Model Description: patients with decompensated cirrhosis with frequent hepatic encephalopathy (HE) or difficult to treat ascites were included if they had chronic active HCV
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cases (Active Comparator): patients with decompensated cirrhosis
  treated with Sofosbuvir 400 mg (Sovaldi) + Daclatasvir 60mg (Daklinza) + Ribavirin 200 mg (Rebetol)
  Interventions: Drug: Sofosbuvir 400mg (Sovaldi) + Daclatasvir 60 mg (Daklinza) + Ribavirin 200 mg (Rebetol)
- control group (Placebo Comparator): the control group treated with liver support including silymarin 140 + phytomenadione 10 mg + lasilactone 50 mg + albumin infusion
  Interventions: Drug: vitamin K (Phytomenadione) 10 mg+ furosemide and spironolactone (Lasilactone) 50 mg + milk thistle (Silymarin) 140 mg + Albumin infusion

INTERVENTIONS:
Drug: Sofosbuvir 400mg (Sovaldi) + Daclatasvir 60 mg (Daklinza) + Ribavirin 200 mg (Rebetol) — sofosbuvir 400mg+ribavirin 400mg+daclatasvir 60 mg were adminstered for 3 months
  Other Names: Direct Acting Antivirals (DAAs)
  Arms: cases
Drug: vitamin K (Phytomenadione) 10 mg+ furosemide and spironolactone (Lasilactone) 50 mg + milk thistle (Silymarin) 140 mg + Albumin infusion — symptomatic therapy for liver support, control of ascites and bleeding tendency.
  Other Names: liver support therapy
  Arms: control group

SUMMARY:
-The limited treatment varieties of decompensated cirrhosis due to hepatitis C virus (HCV) remain a challenge. In patients with reduced hepatic reserve, DAAs may be associated with complications as worsening decompensation. The impact of DAAs therapy on mortality in decompensated cirrhosis was not investigated.

DETAILED DESCRIPTION:
An observational case-control study which was conducted from June 2015 till the first of January 2018 in the Hepatology clinic - Zagazig University hospital-Egypt which is a tertiary referral center.

Out of 422 patients presented with decompensated cirrhosis due to HCV, 342 patients were excluded due to Hepatocellular carcinoma (n=61), cirrhotic cardiomyopathy (n=21), renal impairment (n=34), ischemic heart disease (n=37), active gastrointestinal bleeding (n=42), avoided treatment with DAAs and preferred conservative therapy (n=147); finally 80 patients with decompensated cirrhosis who were willing to be treated and showed frequent hepatic encephalopathy (HE) or difficult to treat ascites were selected to receive DAAs and included if they had chronic HCV proved by the positivity of HCV RNA and elevated transaminases. Their CTP score was >9, MELD score was <29 Patients were excluded if they had compensated cirrhosis or HCV without cirrhosis; exposure to previous antiviral therapy; hepatocellular carcinoma; other causes of liver diseases or mixed causes as excessive alcohol consumption, autoimmune liver disease; previous liver transplantation; patients with risk factors of myocardial dysfunction as abnormal T wave in electrocardiogram, ejection fraction (EF) less than 50%, left ventricular ejection fraction (LVEF) less than 50%.

The control group included 80 patients; they sought medical care at the Hepatology outpatient clinic-Zagazig University hospital. They had decompensated liver disease and preferred to be managed conservatively; they desired to avoid treatment by DAAs by themselves (n=43) or by their relatives (n=37) as they were concerned about the potential risk of liver cancer after direct antiviral agents. They were age, sex, CTP and MELD scores matched with the same inclusion and exclusion criteria and had been chosen from the patients who refused the treatment with DAAs (n=147) after their consent to participate in the study, while the remaining patients refused to be enrolled (n=67).

B-Baseline laboratory investigation

* Investigations preliminary to antiviral therapy as liver function tests, Prothrombin time, Prothrombin concentration (%), kidney function tests, complete Blood Count, fasting blood sugar, HBA1c if diabetes was present and serum AFP. For each patient, CTP and MELD scores were calculated.
* Quantitative assessment of HCV load in the serum by real-time Quantitative PCR (COBAS Ampliprep/Taqman HCV monitor version 2.0, with a detection limit of 15 IU/ml; Roche Diagnostic Systems, just before the study in both groups and after the first month, at the end of treatment and 3 months post-treatment to detect SVR 12th in DAAs treated group
* Genotyping for HCV using INNO-LiPA II, based on genotype-specific oligonucleotides from the 5' UTR that are immobilized on a nitrocellulose strip. The probe reactivity patterns were interpreted according to the manufacturer instructions.

C- Abdominal Ultrasonography (USG) The patients were evaluated for criteria of decompensated cirrhosis including shrunken cirrhotic liver and ascites, patients with HCC were excluded. Criteria of portal hypertension as portal vein diameter > 13mm or cavernous transformation, splenic bipolar diameter >13 cm, splenic vein diameter >8 mm or the presence of splenic collaterals. After treatment termination; USG was done every 6 months for a period of 20 months for early detection of HCC or worsening of hepatic decompensation.

D- Treatment exposure and outcome

* Medications The study patients will be given Sofosbuvir 400mg, ribavirin 400mg, and daclatasvir 60 mg for 3 months and will be evaluated for the development of sustained virological response (SVR), the occurrence of complications after DAAs and the effects of SVR on the frequency of hepatic encephalopathy, improvement in ascites control or difficult to treat ascites defined as ascites that rapidly recurs after paracentesis or cannot be completely mobilized despite maximal medications (sodium restriction of less than 2 g/day with maximal dose of furosemide (160 mg) or spironolactone (400 mg) or inability to reach maximum diuretic dose due to emergence of side effects, and after confirming compliance with sodium restrictions if the 24-hour urine sodium level is <78 mEq, also the impact of therapy on Survival.
* Monitoring
* All the patients will have regular biweekly visits in the first 6 months then every 2 months for 20 months. Every visit a full history taking, laboratory evaluation which included complete blood count (CBC), serum creatinine, total and direct bilirubin, serum albumin, serum transaminases, coagulation profile and AFP.

The patients who did not complete the follow-up will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* chronic active HCV proved by the positivity of HCV RNA, elevated transaminases.
* CTP score was >9, MELD score was <29
* Decompensated cirrhosis with frequent hepatic encephalopathy (HE) or difficult to treat ascites

Exclusion Criteria:

* exposure to previous antiviral therapy
* hepatocellular carcinoma
* other causes of liver diseases or mixed causes (excessive alcohol consumption, autoimmune liver disease)
* previous liver transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-05-24 (Actual); Study Completion 2018-06-24 (Actual)

PRIMARY OUTCOMES:
sustained virological response | 3 months after 3 months after treatment termination
  undetectable HCV RNA 3 months after treatment termination by Polymerase Chain Reaction

SECONDARY OUTCOMES:
improved liver synthetic function | 24 months
  improvement of serum albumin
improved liver synthetic function | 24 months
  improvement of coagulation profile
improved liver excretory function | 24 hours
  improvement of serum total bilirubin

CONTACTS AND LOCATIONS:
Overall Officials: Amr S Hanafy, md, Principal Investigator — Assistant prof of medicine-Zagazig University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hanafy AS, Bassiony MA, Basha MAA. Management of HCV-related decompensated cirrhosis with direct-acting antiviral agents: who should be treated? Hepatol Int. 2019 Mar;13(2):165-172. doi: 10.1007/s12072-019-09933-8. Epub 2019 Feb 13. PMID 30758786